CLINICAL TRIAL: NCT05354336
Title: A Randomized, Open-Label, Phase I Clinical Study on SHR6390 of Different Specifications After Process Modification in Healthy Chinese Volunteers
Brief Title: A Phase I Clinical Study on SHR6390 in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR6390-I-105
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR6390（100mg） (Experimental)
  Interventions: Drug: SHR6390(100mg)
- SHR6390（125mg） (Experimental)
  Interventions: Drug: SHR6390(125mg)
- SHR6390（150mg） (Experimental)
  Interventions: Drug: SHR6390(150mg)

INTERVENTIONS:
Drug: SHR6390(100mg) — SHR6390 at a single oral dose of 100 mg.
  Arms: SHR6390（100mg）
Drug: SHR6390(125mg) — SHR6390 at a single oral dose of 125 mg.
  Arms: SHR6390（125mg）
Drug: SHR6390(150mg) — SHR6390 at a single oral dose of 150 mg.
  Arms: SHR6390（150mg）

SUMMARY:
This study was to evaluate the pharmacokinetics and safety of SHR6390 at doses of 100 mg, 125 mg, and 150 mg after process modification in Chinese healthy volunteers. A single oral dose of SHR6390 was given to each group, including 100 mg, 125mg and 150mg of SHR6390.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese male and female aged 18-45years with a minimum weight of 50 kg for male and 45 kg for female subjects and a body mass index (BMI) of 18-26 kg/m2 who provided written informed consent for participating in the study.
* Without history of cardiovascular, hepatic, kidney, pulmonary, endocrine, gastrointestinal, neurological, or psychiatric disease.
* No pregnancy plan during the trial or within 6 months after completion of the trial.
* Voluntarily signed the informed consent form and strictly adherence to the study protocol.

Exclusion Criteria:

* vital signs, physical examination, 12-lead electrocardiogram, and laboratory examination had results of clinical significance.
* Hepatitis B and C, human immunodeficiency virus (HIV) and syphilis antibody positive;
* Any history of allergy, alcohol and drug abuse;
* blood donation, massive blood loss (≥400mL).
* Participated in other clinical trials within three months. (6) Severe infection or surgery four weeks prior to screening;
* use of any drug that inhibits or induces hepatic metabolizing enzymes four weeks prior to screening;
* use of any prescription drugs, over-the-counter drugs, Chinese herbal medicines and health care products fourteen days prior to screening;
* A history of dysphagia, gastrointestinal ulcers, or any gastrointestinal disease that interferes with drug absorption.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — half male and half female
Enrollment: 36 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2019-08-24 (Actual); Study Completion 2019-08-24 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 12 days
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC)0-t | 12 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-t
Area under the plasma concentration versus time curve (AUC)0-∞ | 12 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-∞

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 22 days
  Collection of adverse events
Incidence of abnormal blood pressure | 22 days
  Monitor both systolic and diastolic blood pressure
Incidence of abnormal temperature | 22 days
  Monitor the temperature
Incidence of abnormal electrocardiogram waveform | 22 days
  Electrocardiogram inspection

CONTACTS AND LOCATIONS:
Locations (1):
- Phase I Clinical Research Center, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No